CLINICAL TRIAL: NCT00783562
Title: Effectiveness of an Extension-Oriented Exercise Program in Preventing Neck and Low Back Complaints in Nursery School Teachers
Brief Title: Preventive Intervention in Nursery School Teachers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Paolo Pillastrini, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PP001032008
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Low Back Pain; Neck Pain
Keywords: Low back pain; Neck pain; Functional disability; Nursery school teachers; Exercise program; Prevention
MeSH Terms: conditions — Low Back Pain; Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: Extension-oriented exercise program; Other: Informative Brochure
- 2 (Active Comparator)
  Interventions: Other: Informative Brochure

INTERVENTIONS:
Other: Extension-oriented exercise program — The exercise program was composed of six graded sessions, two per week for three consecutive weeks. Sessions, each of one hour length, were conducted after the working hours in a wide room of the nursery school, gathering together all the teachers from each school. The exercises were selected in order to reinforce lumbar extension and to strengthen the primary stabilizers of the spine (transversus abdominis, oblique abdominal, multifidus, quadratus lumborum and erector spinae muscles)
  Other Names: EOTA
  Arms: 1
Other: Informative Brochure — The brochure showed the correct way to lift loads, and provided ergonomic suggestions to prevent musculoskeletal complaints, according to the Italian legislation
  Other Names: Educational; Informative Pamphlet

SUMMARY:
Childcare in nursery schools has been shown to be associated with an elevated prevalence of neck, shoulder, arm and low back disorders. The current evidence suggests that exercises seem to be the only effective preventive intervention. Thus the purpose of this study is to determine the effectiveness of an extension-oriented exercise program in preventing low back/neck pain and functional disability in nursery school teachers. In addition, the investigators also sought to identify the occurrence of musculoskeletal complaints in this category of workers.

DETAILED DESCRIPTION:
Seventy-one nursery school teachers working in nine school buildings were randomly divided into two groups, with each school as a unit of randomization. All the teachers in both groups received an ergonomic brochure; teachers in the experimental group also received an extension-oriented exercise program, conducted by a physical therapist. Data were collected at baseline and at a two-month follow-up. The primary outcome measure recorded was the level of disability (Roland Morris Disability Questionnaire and Oswestry Disability Index), while secondary outcome measures included LBP and neck pain presence (Pain Drawing) and intensity (Visual Analogue Scale). At follow-up, a significant improvement was registered in the experimental group for all the outcomes evaluated. In conclusion a six-session extension-oriented exercise program proved decisive in preventing low back and neck complaints and in reducing consequent LBP functional disability among nursery school teachers.

ELIGIBILITY:
Inclusion Criteria:

The study population was composed by all the 71 nursery school teachers, employed at the town hall of Forlì, that worked in nine different school buildings similar in size and furniture. As provided for by the Italian law (Emilia-Romagna Regional Law No. 1 of January 10, 2000 - art. 32, followed by the Directive of July 25, 2001), teachers had the same working schedule and the same workload in terms of teacher/children ratio depending on children age.

Exclusion Criteria:

* medical history of serious injury
* spinal surgery
* malignant pathology

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire and Oswestry Disability Index | Baseline, 2 months

SECONDARY OUTCOMES:
Pain Drawing and Visual Analogue Scale | Baseline, 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, MSc, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Result] Browder DA, Childs JD, Cleland JA, Fritz JM. Effectiveness of an extension-oriented treatment approach in a subgroup of subjects with low back pain: a randomized clinical trial. Phys Ther. 2007 Dec;87(12):1608-18; discussion 1577-9. doi: 10.2522/ptj.20060297. Epub 2007 Sep 25. PMID 17895350
- [Result] Grant KA, Habes DJ, Tepper AL. Work activities and musculoskeletal complaints among preschool workers. Appl Ergon. 1995 Dec;26(6):405-10. doi: 10.1016/0003-6870(95)00057-7. PMID 15677041
- [Result] Brown MZ, Gerberich SG. Disabling injuries to childcare workers in Minnesota, 1985 to 1990. An analysis of potential risk factors. J Occup Med. 1993 Dec;35(12):1236-43. PMID 8113928